CLINICAL TRIAL: NCT04960501
Title: Comparison of Curative Effect Between New Tension Band and Patellar Tension Reduction Band in the Treatment of Lower Pole Fractures of Patella
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUTH ZHS PF
Record Dates: First submitted 2021-07-02; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Follow-up Time, Postoperative Knee Joint Score, Postoperative X-ray, Follow-up Postural Image Data

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New tension band system
  Interventions: Procedure: New type of tension band or patellar tension reduction band for treatment of lower pole fracture of patella
- Patella reduction band system
  Interventions: Procedure: New type of tension band or patellar tension reduction band for treatment of lower pole fracture of patella

INTERVENTIONS:
Procedure: New type of tension band or patellar tension reduction band for treatment of lower pole fracture of patella — New type of tension band or patellar tension reduction band for treatment of lower pole fracture of patella

SUMMARY:
Research purposes:

Analyze the curative effect of the new tension band system composed of φ3.0mm hollow nails, titanium cables and new gaskets and the patellar tension reduction band in the treatment of lower pole fractures of the patella.

research method: A retrospective study of 41 cases of comminuted fractures of the lower pole of the patella treated with a new tension band system composed of φ3.0mm hollow nails, titanium cables and new spacers from March 2012 to July 2017, including 19 males and 22 females , The average age is 56.7 years (22 to 79 years), 24 cases of AO/OTA A1 type, and 17 cases of C1.3 type. During the same period, 22 cases of comminuted fractures of the lower pole of the patella were treated with a patella tension band, including 8 males and 14 females, with an average age of 57.4 years (32 to 84 years), 17 cases of AO/OTA type A1, and 5 cases of type C1.3. The injury mechanism is all slipping and kneeling injuries.

DETAILED DESCRIPTION:
Research purposes:

Analyze the curative effect of the new tension band system composed of φ3.0mm hollow nails, titanium cables and new gaskets and the patellar tension reduction band in the treatment of lower pole fractures of the patella.

research method: A retrospective study of 41 cases of comminuted fractures of the lower pole of the patella treated with a new tension band system composed of φ3.0mm hollow nails, titanium cables and new spacers from March 2012 to July 2017, including 19 males and 22 females , The average age is 56.7 years (22 to 79 years), 24 cases of AO/OTA A1 type, and 17 cases of C1.3 type. During the same period, 22 cases of comminuted fractures of the lower pole of the patella were treated with a patella tension band, including 8 males and 14 females, with an average age of 57.4 years (32 to 84 years), 17 cases of AO/OTA type A1, and 5 cases of type C1.3. The injury mechanism is all slipping and kneeling injuries.

ELIGIBILITY:
Inclusion Criteria:Patients with comminuted fractures of the lower pole of the patella: AO/OTA type A1 and C1.3 type -

Exclusion Criteria:1. Except for other types of patella fractures 2. Except for open patella fractures 3. Excluding patients with other fractures and injuries 4. Exclude patients who cannot cooperate with functional exercises

-

Ages: 22 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Among them, 19 were males and 22 were females, with an average age of 56.7 years (22 to 79 years)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
operation time | One day after surgery

SECONDARY OUTCOMES:
Surgical bleeding | One day after surgery

OTHER OUTCOMES:
Knee joint score after surgery | One week, one month, three months, six months after operation
Postoperative X-ray | One week, one month, three months, six months after operation
Follow-up body image data | One week, one month, three months, six months after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided